CLINICAL TRIAL: NCT02584530
Title: A Randomized Controlled Trial Comparing Ultrasound Guided PICC Line Insertion in Neonates With Standard Procedure
Brief Title: Comparing Ultrasound Guided PICC Line Insertion in Neonates With Standard Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Nadya Ben Fadel, Neonatologist, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20150456
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Ultrasonography, Interventional; Peripheral Venous Catheterization
Keywords: ultrasound; PICC line; neonate
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard procedure group (No Intervention): PICC line insertion using anatomical landmarks guidance and tip placement confirmation by X-ray
- Interventional group (Experimental): Ultrasound guidance for PICC line placement and X-ray
  Interventions: Procedure: Ultrasound guidance for PICC line placement

INTERVENTIONS:
Procedure: Ultrasound guidance for PICC line placement — Apply ultrasound guidance for PICC line placement and positioning in newborns
  Arms: Interventional group

SUMMARY:
This is a randomized controlled study comparing US guided vs standard procedure for PICC line placement in newborns admitted to Children's Hospital of Eastern Ontario Neonatal Intensive Care Unit who require a PICC line. Patients will be randomized using REDCap randomization module (stratified by gestational age < 28 weeks and >= 28 weeks and blocked to ensure approximate balance with each stratum) into two arms. - Arm 1: PICC line insertion procedure using anatomical landmarks and tip placement will be confirmed by X-ray (current standard); Arm 2: US guided PICC line insertion procedure and tip placement confirmation by both US and X-ray. Sample size of 33 infants per group would achieve greater than 80% power to detect a difference between groups.

Primary outcome: Time to complete the standard versus the US-guided procedure.

Secondary outcomes (comparison between two arms):

The number of total "venipuncture" attempts needed to place a PICC line Number of tip manipulations after complete insertion Proportion of successful tip placement

DETAILED DESCRIPTION:
Background Peripherally Inserted Central Catheter (PICC) line placement is one of the most commonly performed procedures in Neonatology. Due to prematurity and small vein size, the procedure often requires multiple attempts over an increased timeframe. As a standard of care, the position is confirmed by X-ray. Frequently, catheters are not optimally positioned, necessitating repositioning and further radiographs.

The use of ultrasound (US) guidance for PICC line placement enhances the visualization of the veins and provides a better selection for optimal access. It could decrease or even eliminate the need for X-rays when used to confirm the tip position.

Objectives To demonstrate that using US-guidance to place and confirm tip positioning for PICC line insertion in neonates will decrease the number of cannulation attempts, will shorten the time needed to complete the procedure, and will decrease infants' exposure to radiation.

Methods This is a randomized controlled study comparing US guided vs standard procedure for PICC line placement in newborns admitted to CHEO NICU who require a PICC line (approximately 130-150 infants per year). Patients will be randomized using REDCap randomization module (stratified by gestational age < 28 weeks and >= 28 weeks and blocked to ensure approximate balance with each stratum) into two arms - Arm 1: PICC line insertion procedure using anatomical landmarks and tip placement will be confirmed by X-ray (current standard); Arm 2: US guided PICC line insertion procedure and tip placement confirmation by both US and X-ray. A sample size of 33 infants per group would be sufficient to achieve greater than 80% power to detect a difference between groups.

Results of this study may demonstrate that US guided PICC line placement is superior (shorter and safer procedure, reduced radiation and pain) to currently used procedure and could lead to practice change.

ELIGIBILITY:
Inclusion Criteria:

All newborns (0-28 days) admitted to Neonatal Intensive Care Unit who require PICC line insertion after consent has been obtained to include in this study. Including:

* Infants who need prolonged Total Parenteral Nutrition requirement of > 7 days.
* Infants with difficult peripheral venous access who requires a central line
* Infants who require IV medications for > 7 days.
* Infants who require medications given by central IV access
* Infants who will undergo complex surgical procedures and will require central IV access before procedure.

Exclusion Criteria:

* Infants requiring isolation according to infection control protocols
* Unable to obtain or refused consent for PICC line and/or study enrolment
* Infants with any clinical contraindication for PICC line insertion as per unit policy

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Time to complete the standard versus the US-guided procedure | one year
  Comparison between total time of procedure with standard approach vs US guidance measured in minutes.

SECONDARY OUTCOMES:
Number of total venipuncture attempts needed to place a PICC line | One year
  Number of venipuncture attempts will be documented per patient through the whole duration of study and then both groups will be compared differences in number
Number of tip manipulations after complete insertion | One year
  Number of manipulations of tip line for adequate placement will be documented on each patient and then compared against control group to assess for differences in number.
Proportion of successful tip placement | One year
  Total number of correct position of PICC line tip will be documented in both groups and then compared to control.

CONTACTS AND LOCATIONS:
Overall Officials: Nadya Ben Fadel, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada